CLINICAL TRIAL: NCT06238895
Title: Optimizing Dosing Strategies in Oral Iron Supplementation
Acronym: OPTIDOSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Helene Meyer, Principal Investigator, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02317
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiencies; Iron Deficiency Anemia; Iron Deficiency Anemia Treatment
Keywords: iron deficiency anemia; oral iron supplementation; iron supplementation; gender differences
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — ferrous sulfate, mucin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Oral iron supplementation with Eisen-II-Sulfat (Tardyferon ®) Every second day 2 x 80 mg Tardyferon® for a duration of 12 weeks.
  Interventions: Drug: Tardyferon
- Active Control (Active Comparator): Oral iron supplementation with Eisen-II-Sulfat (Tardyferon ®) Every day 1x 80 mg Tardyferon® for a duration of 12 weeks
  Interventions: Drug: Tardyferon

INTERVENTIONS:
Drug: Tardyferon — Interval Dosing Strategy (Administration of oral iron every second day with double the standard dose instead of every day standard dose)

SUMMARY:
The goal of this clinical trial is to evaluate, if a change in dosing strategy in oral iron supplementation from leads to an improvement of iron absorption and consequently a faster therapy in patients with iron deficiency.

The main question the study aims to answer is: Does a treatment effect (measured by change in hemoglobin after 12 weeks of treatment) exist between daily oral iron supplementation and interval administration (every second day)? Participants will receive oral iron supplementation every second day with double the standard dose (intervention group). Researchers will compare this group with the active control group, that receives oral iron supplementation every day with the standard dose.

Participants will present for three patient visits (at baseline, after 6 and after 12 weeks of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* ≥18 years of age
* Iron deficiency: Ferritin <30 µg/l
* hemoglobin ≥ 80 g/l
* CRP < 5 mg/l

Exclusion Criteria:

* Refusal of study participation,
* Regular administration of Erythropoietin
* Oral or intravenous iron supplementation <12 weeks prior to investigation
* Contraindications to intervention medication (Tardyferon), e.g. known hypersensitivity or allergy to iron sulfate / ferrous sulfate
* Blood transfusion or donation <12 weeks prior to investigation
* Active chemotherapy
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject.

Note

Due to slow recruitment, the following inclusion criterion was removed on 09/25/2024 (MM/DD/YYYY):

Anemia (as defined by the WHO): Hemoglobin <130 g/L for men, Hemoglobin <120 g/l for women, Hemoglobin <110 g/l for pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Change of Hemoglobin after 12 weeks | 12 weeks
  Change (from baseline before treatment) of hemoglobin after 12 weeks of oral iron supplementation

SECONDARY OUTCOMES:
Proportion of participants achieving treatment goal | 12 weeks
  Proportion of participants achieving either increase of hemoglobin (>20 g/l), normalization of hemoglobin (women >120 g/l, pregnant women >110 g/l and men >130 g/l) after 12 weeks of oral iron supplementation
Change of iron parameters from baseline | 12 weeks
  Change of iron parameters from baseline compared to after treatment of 12 weeks
Side effects | 12 weeks
  Side effects during treatment with oral iron supplementation in both groups (intervention and active control)

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No